CLINICAL TRIAL: NCT00882947
Title: Post-Marketing Surveillance of Ventavis® in Chinese Patients With Primary Pulmonary Hypertension (PPH)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Schering Pharma AG
Other Study IDs: 14183; VE0611CN
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Primary Hypertension
Keywords: Primary Pulmonary Hypertension (PPH)
MeSH Terms: conditions — Essential Hypertension; Familial Primary Pulmonary Hypertension | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Ventavis (Iloprost, BAYQ6256)

INTERVENTIONS:
Drug: Ventavis (Iloprost, BAYQ6256) — Iloprost solution for inhalation, BAYQ6256, Synthetic Prostacyclin analog

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of inhaled Iloprost (Ventavis®) among adult Chinese patients with primary pulmonary hypertension, which is in compliance with Chinese SFDA regulation.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female age 18-65 years old
* The treating physician has chosen Ventavis as a suitable long-term treatment for the patient
* Patient with Primary Pulmonary Hypertension (i.e. IPAH or FPAH) and classified as NYHA functional class III
* Written informed/data protection consent
* No prior treatment with Ventavis or other active treatments for PPH within 6 weeks of date of study.

Exclusion Criteria:

* Known or newly identified contraindication for administration of Ventavis as stated in the Ventavis product package insert.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Chinese patients (age 18-65 male and female) with Primary Pulmonary Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2006-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | At week 4,12 and 24

SECONDARY OUTCOMES:
6 minute walking test (6-MWT) | At week 4,12 and 24
NYHA functional class | At week 4,12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China